CLINICAL TRIAL: NCT02651922
Title: Treatment of Patients Suffering From Nervous Restlessness With PASCOFLAIR®
Status: Completed | Type: Observational
Sponsor: Pascoe Pharmazeutische Praeparate GmbH (Industry)
Collaborators: Institut für Empirische Gesundheitsökonomie, Prof. Dr. Dr.med. Reinhard Rychlik,Am Ziegelfeld 28,51399 Burscheid,Germany (Unknown)
Responsible Party: Sponsor
Other Study IDs: 199A14PF
Record Dates: First submitted 2016-01-06; First posted 2016-01-11 (Estimated); Results first posted 2017-06-19 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Nervous Restlessness
Keywords: Nervous restlessness; Pascoflair; Passiflora incarnata; Benzodiazepine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The study was carried out as a prospective, non-interventional study with the intention of subsequent process cost analyses (PCA) and also considers quality of life, drug misuse, dependence, adverse events and therapy satisfaction.

DETAILED DESCRIPTION:
The study was carried out as a prospective, non-interventional study with the intention of subsequent process cost analyses (PCA) and also considers quality of life, drug misuse, dependence, adverse events and therapy satisfaction. Data were collected in collaboration with 22 physicians in Germany.

The study was designed as a one armed non-interventional study. Patients had to suffer from nervous restlessness in order to be eligible for study documentation. Participants agreed to a medical treatment with PASCOFLAIR® of 12 weeks. In this context, documented patients could take PASCOFLAIR® at the first time or could have started within the past three months before the initial visit. Furthermore, documented patients had to be older than 18 years and must be able to read and understand the patient declaration of data protection and the declaration of consent. The patient must not be an alcoholic, must not be drug dependent and have no other types of addiction. Patients who were pregnant or breast-feeding were not eligible for study participation. Furthermore, patients showing hypersensitivity against passionflower extract or against other components of the medication were excluded. The signed declaration of consent of participating patients is available.

The treatment of affected patients may not be documented, if a redemption (written or spoken) of the declaration of consent is existing or the patient takes Benzodiazepines.

ELIGIBILITY:
Inclusion Criteria:

* patients suffering from nervous restlessness

Exclusion Criteria:

* Age < 18 years and must be able to read and understand the patient declaration of data protection and the declaration of consent
* alcoholics, drug pending, addictive disorder
* pregnancy or lactating
* patients showing hypersensitivity against passionflower extract or against other components of the medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients had to suffer from nervous restlessness in order to be eligible for study documentation.
Sampling Method: Probability Sample
Enrollment: 154 (Actual)
Dates: Start 2014-09; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- PASCOFLAIR Group (Verum): Patients who were treated with PASCOFLAIR
Period: Overall Study
Arm/Group | PASCOFLAIR Group (Verum)
Started | 156
Completed | 154
Not Completed | 2
Not completed — due to exclusion criteria | 2

BASELINE CHARACTERISTICS:
Population: A total of 156 patients participated in the study. Two patients were excluded from the analysis, because they received Benzodiazepines (Tavor, Lexostad). One patient was 17 years of age when documented in the study. The overall study population considered in the analyses was 154 patients.
Arm/Group | PASCOFLAIR Group (Verum)
Number analyzed (Participants) | 154
Age, Customized [Number; unit: participants] — 2 missinig data
  participants
    <=18 years | 1
    Between 18 and 65 years | 128
    >=65 years | 23
    missing data | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.9 (17.1)
Sex/Gender, Customized [Number; unit: participants]
  Female | 115
  Male | 38
  missing data | 1
Region of Enrollment [Number; unit: participants]
  Germany | 154

OUTCOME MEASURES:

1. Primary Outcome: Change of Symptom Inner Restlessness (Pre - Post)
Description: Symptom was assessed in a Likert scale ranging from 0 "no symptoms at all" to 10 "very severe symptoms"
Time Frame: Change from Baseline (before treatment; week 0) to last visit (end of observation- approx. 12 weeks after baseline)
Population: If a symptom was rated 0, it was considered nonexistent. For any other rating (1 to 10) the symptom was considered existent.
  Only 146 patients showed this symptom.
Measure: Number; unit: participants
Arm/Group | PASCOFLAIR Group (Verum)
Number analyzed (Participants) | 146
participants
  improved | 137
  unchanged | 3
  detoriated | 6

2. Secondary Outcome: Change of Symptom Sleep Disturbance (Pre - Post)
Description: Symptom was assessed in a Likert scale ranging from 0 "no symptoms at all" to 10 "very severe symptoms"
Time Frame: Change from Baseline (before treatment; week 0) to last visit (end of observation- approx. 12 weeks after baseline)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | PASCOFLAIR Group (Verum)
Number analyzed (Participants) | 146
participants
  improved | 131
  unchanged | 8
  deteriorated | 7

3. Secondary Outcome: Change of Symptom Exhaustion (Pre - Post)
Description: Symptom was assessed in a Likert scale ranging from 0 "no symptoms at all" to 10 "very severe symptoms"
Time Frame: Change from Baseline (before treatment; week 0) to last visit (end of observation- approx. 12 weeks after baseline)
Population: If a symptom was rated 0, it was considered nonexistent. For any other rating (1 to 10) the symptom was considered existent.
  Only 145 patients showed this symptom.
Measure: Number; unit: participants
Arm/Group | PASCOFLAIR Group (Verum)
Number analyzed (Participants) | 145
participants
  improved | 130
  unchanged | 7
  detoriorated | 8

4. Secondary Outcome: Change of Symptom Fear (Pre - Post)
Description: Symptom was assessed in a Likert scale ranging from 0 "no symptoms at all" to 10 "very severe symptoms"
Time Frame: Change from Baseline (before treatment; week 0) to last visit (end of observation- approx. 12 weeks after baseline)
Population: If a symptom was rated 0, it was considered nonexistent. For any other rating (1 to 10) the symptom was considered existent.
  Only 133 patients showed this symptom.
Measure: Number; unit: participants
Arm/Group | PASCOFLAIR Group (Verum)
Number analyzed (Participants) | 133
participants
  improved | 121
  unchanged | 6
  detoriorated | 10

5. Secondary Outcome: Change of Symptom Lack of Concentration (Pre - Post)
Description: Symptom was assessed in a Likert scale ranging from 0 "no symptoms at all" to 10 "very severe symptoms"
Time Frame: Change from Baseline (before treatment; week 0) to last visit (end of observation- approx. 12 weeks after baseline)
Population: If a symptom was rated 0, it was considered nonexistent. For any other rating (1 to 10) the symptom was considered existent.
  Only 142 patients showed this symptom.
Measure: Number; unit: participants
Arm/Group | PASCOFLAIR Group (Verum)
Number analyzed (Participants) | 142
participants
  improved | 123
  unchanged | 11
  detoriorated | 8

6. Secondary Outcome: Change of Symptom Transpiration (Pre - Post)
Description: Symptom was assessed in a Likert scale ranging from 0 "no symptoms at all" to 10 "very severe symptoms"
Time Frame: Change from Baseline (before treatment; week 0) to last visit (end of observation- approx. 12 weeks after baseline )
Population: If a symptom was rated 0, it was considered nonexistent. For any other rating (1 to 10) the symptom was considered existent.
  Only 121 patients showed this symptom.
Measure: Number; unit: participants
Arm/Group | PASCOFLAIR Group (Verum)
Number analyzed (Participants) | 121
participants
  improved | 106
  unchanged | 9
  detoriorated | 6

7. Secondary Outcome: Change of Symptom Nausea (Pre - Post)
Description: Symptom was assessed in a Likert scale ranging from 0 "no symptoms at all" to 10 "very severe symptoms"
Time Frame: Change from Baseline (before treatment; week 0) to last visit (end of observation-approx. 12 weeks after baseline)
Population: If a symptom was rated 0, it was considered nonexistent. For any other rating (1 to 10) the symptom was considered existent.
  Only 92 patients showed this symptom.
Measure: Number; unit: participants
Arm/Group | PASCOFLAIR Group (Verum)
Number analyzed (Participants) | 92
participants
  improved | 79
  unchnaged | 7
  detoriorated | 6

8. Secondary Outcome: Change of Symptom Trembling (Pre - Post)
Description: Symptom was assessed in a Likert scale ranging from 0 "no symptoms at all" to 10 "very severe symptoms"
Time Frame: Change from Baseline (before treatment; week 0) to last visit (end of observation - approx. 12 weeks after baseline)
Population: If a symptom was rated 0, it was considered nonexistent. For any other rating (1 to 10) the symptom was considered existent.
  Only 108 patients showed this symptom.
Measure: Number; unit: participants
Arm/Group | PASCOFLAIR Group (Verum)
Number analyzed (Participants) | 108
participants
  improved | 91
  unchanged | 8
  deterioreated | 9

9. Secondary Outcome: Change of Symptom Palpation (Pre - Post)
Description: Symptom was assessed in a Likert scale ranging from 0 "no symptoms at all" to 10 "very severe symptoms"
Time Frame: Change from Baseline (before treatment; week 0) to last visit (end of observation- approx. 12 weeks after baseline)
Population: If a symptom was rated 0, it was considered nonexistent. For any other rating (1 to 10) the symptom was considered existent.
  Only 130 patients showed this symptom.
Measure: Number; unit: participants
Arm/Group | PASCOFLAIR Group (Verum)
Number analyzed (Participants) | 130
participants
  improved | 117
  unchanged | 9
  deteriorated | 4

10. Secondary Outcome: Change of BDEPQ (Benzodiazepine Dependence Questionnaire)
Description: The Benzodiazepine Dependence Questionnaire (BDEPQ) is a 30 item self report questionnaire designed to measure dependence on benzodiazepine tranquilisers, sedatives and hypnotics. Items cover all aspects of the dependence syndrome with the exception of withdrawal symptoms. Each item is rated on a four point likert scale referring to experiences in the last month.
  BDEPQ score ranges from 0 (no dependence) to 85 (most severe dependence).
Time Frame: Change from visit 2 (approx. 4 weeks after baseline) to last visit (end of observation- approx. 12 weeks after baseline)
Population: For patient with less than 75% items answered the BDEPQ-Score was not calculated.
  For only 132 patients Score was calculated.
Measure: Number; unit: participants
Arm/Group | PASCOFLAIR Group (Verum)
Number analyzed (Participants) | 132
participants
  improved | 91
  unchanged | 13
  deteriorated | 28

11. Secondary Outcome: Change of RS-13 (Resilience Questionnaire) (Pre - Post)
Description: RS-13 is a 13 items self Report questionnaire measure the resilience, which applies a reliance scale ranging from 13 (lowest stress resistance) to 91 (highest stress resistance).
Time Frame: Change from Baseline (before treatment; week 0) to last visit (end of observation- approx. 12 weeks after baseline)
Measure: Number; unit: participants
Arm/Group | PASCOFLAIR Group (Verum)
Number analyzed (Participants) | 132
participants
  improved | 115
  unchanged | 3
  deteriorated | 14

12. Secondary Outcome: Change in EQ-5D (Health Questionnaire) Scores (Pre - Post)
Description: EQ-5D™ is a standardised instrument for use as a measure of health Outcome The EQ-5D assesses five aspects of QoL: mobility, self-care, usual activity, pain/discomfort and anxiety/depression. An EQ-5D profile score of 0 points represents the worst QoL (death), while 1 point stands for full health. Data analysis was performed according to the EuroQol manual. The EQ-VAS ranges from 0 (worst QoL) to 100 (best QoL).
Time Frame: Change from Baseline (before treatment) to last visit (end of observation- approx. 12 weeks after baseline)
Measure: Number; unit: participants
Arm/Group | PASCOFLAIR Group (Verum)
Number analyzed (Participants) | 133
participants
  improved | 104
  unchanged | 22
  deterioreated | 7

13. Secondary Outcome: Change of EQ-5D VAS Scores (Pre - Post)
Description: VAS values (Quality of Life) range from 0 (very poor) to 100 (best possible state).
Time Frame: Change from Baseline (before treatment; week 0) to last visit (end of observation- approx. 12 weeks after baseline)
Measure: Number; unit: participants
Arm/Group | PASCOFLAIR Group (Verum)
Number analyzed (Participants) | 134
participants
  improved | 119
  unchanged | 5
  deteriorated | 11

14. Secondary Outcome: Tolerability Assess Using a 5 Point Scale
Description: Assessment of tolerability using a 5 point scale (very good, good, satisfactory, bad, very bad)
Time Frame: Evaluation of Tolerability on visit 3 (appr. 12 weeks after baseline)
Measure: Number; unit: participants
Arm/Group | PASCOFLAIR Group (Verum)
Number analyzed (Participants) | 148
participants
  very good | 109
  good | 35
  satisfactory | 2
  bad | 1
  very bad | 1

ADVERSE EVENTS:
Time Frame: The observational period was from September 2014 till June 2015. Per Patient were adrs collected for the treatment period (12 weeks).
Arm/Group | PASCOFLAIR Group (Verum)
Serious Adverse Events (participants affected / at risk) | 0/154
Other Adverse Events (participants affected / at risk) | 3/154
OTHER ADVERSE EVENTS (reported when occurring in more than 1.0% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PASCOFLAIR Group (Verum) (N=154)
Fatigue (Gastrointestinal disorders) | 3 (3)
Numbness in limbs (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No